CLINICAL TRIAL: NCT01869166
Title: Clinical Study of Chimeric EGFR Antigen Receptor-modified T Cells in Chemotherapy Refractory Advanced Solid Tumors
Brief Title: Treatment of Chemotherapy Refractory EGFR(Epidermal Growth Factor Receptor) Positive Advanced Solid Tumors (CART-EGFR)
Acronym: CART-EGFR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor and Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-007
Record Dates: First submitted 2013-06-01; First posted 2013-06-05 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Advanced EGFR-positive Solid Tumors
Keywords: chemotherapy and/or EGFR-antibody/kinase inhibitor therapy refractory solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-tumor response of CART-EGFR (Experimental)
  Interventions: Biological: CART-EGFR

INTERVENTIONS:
Biological: CART-EGFR

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is to study genetically engineered lymphocyte therapy in treating patients with EGFR positive advanced/unresectable operation solid tumors, such as lung cancer, colorectal cancer，ovary cancer，cholangiocarcinoma，pancreatic cancer，renal carcinoma and other relapsed/metastatic tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-EGFR Lentivirus vector (referred to as CART-EGFR cells).

II. Determine duration of in vivo survival of CART-EGFR cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of CART-EGFR CD3zeta:CD137 over time.

SECONDARY OBJECTIVES:

I. For patients with advanced， relapsed/metastatic cancers, measure anti-tumor response due to CART-EGFR cell infusions.

II. Estimate relative trafficking of CART-EGFR cells in tumor bed.

III. Determine if cellular or humoral host immunity develops against the murine anti-EGFR, and assess correlation with loss of detectable CART-EGFR (loss of engraftment).

IV. Determine the relative subsets of CART-EGFR T cells (Tcm, Tem, and Treg).

OUTLINE: Patients are assigned to 1 group according to order of enrollment.

Patients receive anti-EGFR-CAR (coupled with CD137 and CD3 zeta signalling domains)Lentivirus vector-transduced autologous T cells for 3-5 days in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

Estimate relative trafficking of CART-EGFR cells in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Chemotherapy refractory EGFR-positive non-small cell lung cancer, colorectal cancer with liver metastasis,and chemotherapy resistant or relapsed ovary cancerlung cancer,cholangiocarcinoma，pancreatic cancer，renal carcinoma and other relapsed/metastatic/unresectable operation tumors.the expression of EGFR in tumor is more than 50%.
2. Relapsed patients after anti-EGFR using antibody or kinase inhibitor therapy.
3. Patients must be 18 years of age or older.
4. Patients must have an ECOG (Eastern Cooperative Oncology Group )performance status of 0-2.
5. Patients must have evidence of adequate hepatic and renal function as evidenced by the following laboratory parameters:

   Absolute neutrophil count greater than 1500/mm3. Platelet count greater than 100,000/mm3. Hemoglobin greater than 10g/dl (patients may receive transfusions to meet this parameter).

   Total bilirubin < 1.5 times upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).
6. Seronegative for HIV antibody.
7. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody.
8. Patients must be willing to practice birth control during and for four months following treatment.NOTE:women of child-bearing age must have evidence of negative pregnancy test.
9. Patients must be willing to sign an informed consent.

Exclusion Criteria:

1. Patients with life expectancy less than 12 months will be excluded.
2. Patients with uncontrolled hypertension (> 160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months of study will be excluded.
3. Patients with any of the following pulmonary function abnormalities will be excluded: FEV(forced expiratory volume), < 30% predicted; DLCO (diffusing capacity of lung for carbon monoxide) < 30% predicted (post-bronchodilator); Oxygen Saturation less than 90% on room air.
4. Patients with severe liver and kidney dysfunction or consciousness disorders will be excluded.
5. Pregnant and/or lactating women will be excluded.
6. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.
7. Patients with any type of primary immunodeficiencies will be excluded from the study.
8. Patients requiring corticosteroids (other than inhaled) will be excluded.
9. Patients with history of T cell tumors will be excluded.
10. Patients who are participating or participated any other clinical trials in latest 30 days will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24

SECONDARY OUTCOMES:
Anti-tumor responses to CART-EGFR cell infusions | up to 24 weeks

OTHER OUTCOMES:
in vivo existence of CART-EGFR | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: weidong han, Dr., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu Y, Guo Y, Wu Z, Feng K, Tong C, Wang Y, Dai H, Shi F, Yang Q, Han W. Anti-EGFR chimeric antigen receptor-modified T cells in metastatic pancreatic carcinoma: A phase I clinical trial. Cytotherapy. 2020 Oct;22(10):573-580. doi: 10.1016/j.jcyt.2020.04.088. Epub 2020 Jun 9. PMID 32527643
- [Derived] Guo Y, Feng K, Liu Y, Wu Z, Dai H, Yang Q, Wang Y, Jia H, Han W. Phase I Study of Chimeric Antigen Receptor-Modified T Cells in Patients with EGFR-Positive Advanced Biliary Tract Cancers. Clin Cancer Res. 2018 Mar 15;24(6):1277-1286. doi: 10.1158/1078-0432.CCR-17-0432. Epub 2017 Nov 14. PMID 29138340
- [Derived] Feng KC, Guo YL, Liu Y, Dai HR, Wang Y, Lv HY, Huang JH, Yang QM, Han WD. Cocktail treatment with EGFR-specific and CD133-specific chimeric antigen receptor-modified T cells in a patient with advanced cholangiocarcinoma. J Hematol Oncol. 2017 Jan 5;10(1):4. doi: 10.1186/s13045-016-0378-7. PMID 28057014